CLINICAL TRIAL: NCT06865365
Title: Prospective, Randomized, Controlled Trial of Preoperative Use of Saxenda (Liraglutide) Additionally to Common Dietological Measures as Opposed to Dietological Measures Alone
Brief Title: Preoperative Use of Liraglutide Additionally to Common Dietological Measures as Opposed to Dietological Measures Alone
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Daniel Moritz Felsenreich, Professor (Ap. Prof. Priv. Doz. DDr. ), Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2493/2024
Record Dates: First submitted 2025-01-23; First posted 2025-03-07 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Obesity, Adolescent
Keywords: Obesity; Bariatric surgery; metabolic surgery; liraglutide; saxenda; weight loss; surgery risk reduction; excess weight loss
MeSH Terms: conditions — Pediatric Obesity; Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, open
Masking Description: Masking Description
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A - Control Group with only dietological measures (Active Comparator): Patients seeking bariatricsurgery will recieve the standard dietological measures to prepare for bariatric surgery for 6 months
  Interventions: Behavioral: Dietologic measures and lifestyle optimization for weight loss
- Group B - Intervention with additional Liraglutide (Experimental): Patients seeking bariatricsurgery will recieve the standard dietological measures and additional Liraglutide to prepare for bariatric surgery for 6 months
  Interventions: Drug: Liraglutide daily (0.6-3.0mg, highest tolerable dose) additional to dietological measures and lifestyle optimization suggestions

INTERVENTIONS:
Drug: Liraglutide daily (0.6-3.0mg, highest tolerable dose) additional to dietological measures and lifestyle optimization suggestions — Liraglutide daily (0.6-3.0mg, highest tolerable dose) as additional preoperative method for weight loss
  Arms: Group B - Intervention with additional Liraglutide
Behavioral: Dietologic measures and lifestyle optimization for weight loss — all subjects will receive dietary measures and lifestyle opitmization suggestions in order to drop weight preoperatively.
  Arms: Group A - Control Group with only dietological measures

SUMMARY:
The aim of the study is to investigate the effects of preoperative Saxenda (liraglutide). There are two groups, one group receives Saxena in addition to dietary measures when first seeking the operation, one group only diet. The investigator is researching how much additional preoperative weight loss is possible with the drug admitted preoperatively.

DETAILED DESCRIPTION:
The aim of the study is to investigate the effects of preoperative Saxenda (liraglutide). There are two groups, one group receives Saxena in addition to dietary measures, one group only diet. Each group will have a waiting period of 6 months until the operation will be done. The investigator wants to elaborate how much additional preoperative weight loss is possible with the drug. The greater the preoperative weight loss, the lower the risk of the operation.

After one year, the investigator will also check whether the weight loss has been maintained and whether the preoperative Saxenda continues to lose even more weight after the operation.

All patients looking for bariatric surgery with health insurance via Österreichische Gesundheitsklasse and BMI>35kg/m2 will be asked to take part in this study.

Patients with previous bariatric surgeries or contraindications against liraglutide will be excluded from this study.

ELIGIBILITY:
Inclusion Criteria:

- Patients seeking bariatric surgery

* BMI > 35.0 kg/m2
* Health insurance via Österreichische Gesundheitskasse
* Willingness to be assigned to either of the two groups
* Willingness to adhere to preoperative dietological measures
* Follow-up anticipation with blood draws and body weight scans using Secca scale
* Written informed consent

Exclusion Criteria:

* Patients with previous bariatric surgerys

  * Patients aged below 18 years
  * Patients with BMI < 35 kg/m2
  * Patients with psychiatric disorders
  * Patients not willing to adhere to preoperative dietological measures
  * Patients with contraindications against Saxenda
  * Patients who have health insurance other than Österreichische Gesundheitskasse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
% total weight loss | body weight and bmi will be assessed immediately when admission to the study is done as reference value and at at time of operation, which is 6 months after admission to the study, as outcome value
  calculation using ANCOVA, p-value ≤ 0.05 is considered statistically significant

SECONDARY OUTCOMES:
comorbidities | The secondary parameters will be assessed immediately at the time when admission to the study is done for reference and the time of the surgery, which is 6 months after admission, as outcome parameter
  The secondary parameter will be the prevalence of comorbidities (determined via use of pharmacological therapy therefore)
hba1c | The secondary parameters will be assessed immediately when admission to the study is done for reference and the time of the surgery, which is 6 months after admission, as outcome parameter
  The secondary parameter will be hba1c in %
% weight lost after one year | Body weight will be assessed immediately when admission to the study is done and the time of the surgery (=6 months after admission) and 1 year post op (=18 months after admission)
  % of body weight lost 1 year post op

IPD SHARING:
Plan to Share IPD: No